CLINICAL TRIAL: NCT03217994
Title: Efficacy of a 6% Hydrogen Peroxide Tooth Bleaching Agent Without Ligth
Brief Title: Efficacy of a 6% Hydrogen Peroxide Tooth Bleaching Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Profesor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15/001b
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 37.5% gel (Active Comparator): 37.5% gel to bleach teeth
  Interventions: Drug: gel HP
- 6% gel (Experimental): 6% gel to bleach teeth
  Interventions: Drug: gel HP

INTERVENTIONS:
Drug: gel HP — gel of hygrogen peroxide for teeth bleaching

SUMMARY:
The present study investigates whether it is possible to achieve equally satisfactory results between 37.5% hydrogen peroxide gel and 6% gel for teeth bleaching. A prospective, double-blind, randomized clinical trial was carried out. A total of 33 patients were selected from the clinic of the Faculty of Dentistry at the University of Chile. The patients included men and women over 18 years old without prior tooth whitening treatments, tooth decay, or restorations of the upper front teeth. The patients had tooth colors of A3 or less according to the Vita Classical scale, which was determined with a Vita Easy® Shade spectrophotometer. The study was carried out with a "split-mouth" design. One side of each mouth was randomly treated with 37.5% hydrogen peroxide, and the other side was bleached with 6% hydrogen peroxide. Each group received 3 to 12 minutes of treatment with the respective gel applications. Two sessions of bleaching were carried out each week. Color was assessed at 7 different sessions for 3 months. The spectrophotometer was used to measure the total variation of color (ΔE) between the baseline (session 1) and different measurement times (sessions 2-7). We compared ΔE for both agents using the Mann-Whitney test.

DETAILED DESCRIPTION:
2. Materials and methods

2.1. Study design This study was a double-blind, randomized, prospective clinical trial. The study was conducted according to the recommendations of CONSORT (Consolidated Standards of Reporting Trials) while following the principles of the Helsinki Convention.

2.2. Description of the sample 2.2.1. Selection of the sample

A total of 33 patients were selected from the clinic of the Faculty of Dentistry at the University of Chile. The patients had been seeking whitening treatment and volunteered to participate in the study. The selected patients had to meet all the inclusion criteria and signed informed consent forms (appendix 1) adopted by the Ethics Committee of Faculty of Dentistry. The inclusion criteria were the following:

* Age over 18 years (both sexes)
* 6 present upper front teeth
* No caries
* No restorations (anterosuperior group)
* No previous whitening treatments
* Tooth color value of A3 or less (Vita Classical scale), which was determined with a spectrophotometer (Vita Easy Shade® Compact) on the middle third of the vestibular surface of the maxillary lateral incisors

Patients were excluded based on the following criteria:

* Pregnant or nursing mothers
* In pharmacological treatment
* Bruxopatas and patients who reported prior tooth sensitivity
* Previous tooth whitening (either at home or professionally)
* Visible dental cracks, developmental defects (hypoplasias enamel, hipomineralizaciones, etc.), or teeth stained by tetracycline or fluorosis in the anterosuperior group
* Treatment with fixed appliances
* Periodontal disease or cancer
* Presence of non-carious cervical lesions, or endodontics in the anterosuperior group

Patients who experienced any pathologies that prevented them from entering the study (such as caries, periodontal disease, or dental sensitivity) were directed for treatment to the dental clinic of the Faculty of Dentistry of the University of Chile.

2.2.2. Sample size The sample size n was determined based on similar previous studies (Bortolatto et al., 2014; Martin et al., 2015; Fernandez et al., 2016). A minimum n of 25 patients per group was determined. A significance level of 5% was considered at (1-β) 0.80 with a drop-out rate of 5%.

2.2.3. Study location Treatments were carried out at the clinic of the Faculty of Dentistry of the University of Chile. During this period, volunteers were supervised by the researchers.

2.3. Procedure 2.3.1. Determination of study groups The study was carried out with a "split-mouth" design. Bleaching agents (hydrogen peroxide) were randomly assigned to each hemiarcade. The operators (R.H. and M.P.) were unaware of the product being used. To achieve this, automixed syringes from a Polaoffice+ whitening kit were used (SDI Limited, Bayswater, Australia). The syringes contained hydrogen peroxide in the form of thixotropic gel at a concentration determined by the manufacturer and marked properly.

Each gel syringe was re-labeled with a key number depending on the concentration of the agent, which was determined by an operator (G.Z.) who was unaware of the procedures. All color measurements were performed on the upper lateral incisors by different operators from those mentioned (C.A. and C.A.). In one group, the hemiarcade was bleached with 37.5% hydrogen peroxide (Polaoffice + 37.5% SDI Limited, Bayswater, Australia). In the other group, the hemiarcade was bleached using 6% hydrogen peroxide (Polaoffice + 6% SDI Limited, Bayswater, Australia).

2.3.2. Preliminary phase We first verbally explained the procedures to perform and asked each volunteer to read and sign an informed consent form (appendix 1). A clinic card (appendix 2) was completed for each patient. In each case, a heavy silicone matrix (Speedex® Putty) was prepared for both maxillary lateral incisors. These matrices were drilled at the height of the union of the cervical third with the middle third of the vestibular tooth face to standardize the color measurements with the spectrophotometer (Vita Zahnfabrik, Bad Säckingen, Germany). Another reason was to create a perfect fit with the nozzle of the spectrophotometer to help control the passage of light to the measurement site. The color of each upper lateral incisor was measured using the spectrophotometer, which was previously calibrated according to the manufacturer's instructions using arrays of heavy silicone.

2.3.3. Bleaching protocol Two whitening sessions were carried out with intervals of one week. At the beginning of each session, dental prophylaxis was done with a brush at low speed. Stone pumice and water were used in the upper front to remove the layer from the surface of the teeth enamel so that it would not alter the effectiveness of the gels. We used a plastic lip separator, a blue gingival barrier syringe, and light-curing (Polaoffice + SDI Limited, Bayswater, Australia) to protect the soft tissue. We homogeneously applied the different gels on the vestibular surfaces of each hemiarcade. One hemiarcade was treated with 37.5% hydrogen peroxide, and the other was treated with 6% hydrogen peroxide (Polaoffice + SDI Limited, Bayswater, Australia).

The protocol included 3 applications of 12 minutes each. The gels were in full contact with the tooth surface and then were removed between each application with cotton rolls, which were moistened with water and dried carefully. At the end of the third application, we removed the gels, washed off all excess with plenty of water, and removed the gingival barrier.

2.3.4. After bleaching All patients were instructed to avoid consuming foods with a high content of pigments, such as coffee, tea, wine, and beets during the study period.

2.3.5. Controls At the end of the first session, we measured the color of each lateral incisor with the calibrated spectrophotometer. A week later, the same protocol was repeated. The time to control sessions was considered from the last session of whitening.

Figure 3: Measurement times.

2.3.6. Tabulation of data

Data obtained in each period were tabulated according to the three axes of the CIELAB system (L *, a *, and b *). We also calculated ΔE using the Pythagorean theorem as follows (Westland et al., 2003):

ΔE = [(ΔL)2 + (Δa)2 + (Δb)2]1/2

The variation of each parameter in different times was always calculated in relation to the initial values (the color measurement prior to the first session of whitening).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years (both sexes)
* 6 present upper front teeth
* No caries
* No restorations (anterosuperior group)
* No previous whitening treatments
* Tooth color value of A3 or less (Vita Classical scale), which was determined with a spectrophotometer (Vita Easy Shade® Compact) on the middle third of the vestibular surface of the maxillary lateral incisors

Exclusion Criteria:

* Pregnant or nursing mothers
* In pharmacological treatment
* Bruxism and patients who reported prior tooth sensitivity
* Previous tooth whitening (either at home or professionally)
* Visible dental cracks, developmental defects or teeth stained by tetracycline or fluorosis in the anterosuperior group
* Treatment with fixed appliances
* Periodontal disease or cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Efectiveness by color difference ( using the spectrophotometer Vita Easy Shade) | 1 month
  The shade was determined using the obtained parameters L*, a*, and b* by Spectrophotometer . The color alteration after each session was given by the differences between the values obtained at the session and the baseline (∆E). ∆E was calculated using the following formula: ΔE = [(ΔL*)2 + (Δa*)2 + (Δb*)2]1/2 .

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín, Principal Investigator — University of Chile
Locations (1):
- Eduardo Fernandez, Santiago, N/A = Not Applicable, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Estay J, Angel P, Bersezio C, Tonetto M, Jorquera G, Pena M, Fernandez E. The change of teeth color, whiteness variations and its psychosocial and self-perception effects when using low vs. high concentration bleaching gels: a one-year follow-up. BMC Oral Health. 2020 Sep 11;20(1):255. doi: 10.1186/s12903-020-01244-x. PMID 32917192